CLINICAL TRIAL: NCT00867139
Title: A Pilot, Randomized Study Comparing the Safety, Tolerability and Pharmacokinetics of Combination Therapy (Amantadine, Ribavirin, Oseltamivir) Versus Neuraminidase Inhibitor Monotherapy to Influenza Virus Infected Immunocompromised Patients
Brief Title: TCAD vs. Monotherapy for Influenza A in Immunocompromised Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Michael Boeckh, Member, Vaccine and Infectious Disease Division, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2323.00; 6895 (Other: FHCRC/UW CC IRB); NCT00865800 (obsolete NCT alias)
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Influenza
Keywords: Influenza; Immunocompromised; Antiviral
MeSH Terms: conditions — Influenza, Human | interventions — thiazole-4-carboxamide adenine dinucleotide; Amantadine; Ribavirin; Oseltamivir; Zanamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TCAD-Randomized Arm (Experimental): TCAD (amantadine hydrocholoride, ribavirin and oseltamivir phosphate)
  Interventions: Drug: TCAD
- Neuraminidase Monotherapy Arm (Active Comparator): Zanamivir or Oseltamivir
  Interventions: Drug: Zanamivir or Oseltamivir
- TCAD Open Label Arm (Other): TCAD for subjects who cannot tolerate or are ineligible to receive zanamivir
  Interventions: Other: Open label treatment with TCAD

INTERVENTIONS:
Drug: TCAD — TCAD (amantadine hydrocholoride, ribavirin and oseltamivir phosphate)
  Other Names: Symmetrel; Rebetol; Tamiflu
  Arms: TCAD-Randomized Arm
Drug: Zanamivir or Oseltamivir — Zanamivir or Oseltamivir
  Other Names: Relenza; Tamiflu
  Arms: Neuraminidase Monotherapy Arm
Other: Open label treatment with TCAD — TCAD(amantadine hydrocholoride, ribavirin and oseltamivir phosphate)
  Other Names: Symmetrel; Rebetol; Tamiflu
  Arms: TCAD Open Label Arm

SUMMARY:
The purpose of this study is to assess the safety and tolerability of triple combination antiviral drug (TCAD) for use in immunocompromised patients with Influenza A infection, and to gain data on the effectiveness of TCAD

ELIGIBILITY:
Inclusion Criteria:

i. Inclusion criteria for randomized arms (both needed):

1. Age ≥7 years, male or female; AND
2. Influenza infection (i.e. upper respiratory tract infection)

ii. Inclusion criteria for open-label arm (at least one criteria required):

1. Young age (1-6 years) with any influenza severity, proven or probable influenza A (H1N1)(H274Y); OR
2. History of asthma; OR
3. Older age (≥ 7 years), with no asthma; AND

   * moderate to severe influenza; AND/OR
   * failure in randomized study monotherapy arm iii. Inclusion criteria for all subjects:

1. Able to provide informed consent, or for whom consent may be provided by guardian 2. Immunocompromised, as defined by one of the following:

* Recent hematopoietic cell transplantation (HCT) (within 2 years, all conditioning regimens, allogeneic, autologous, syngeneic; after 2 years patients with chronic graft-versus-host disease (GVHD) requiring systemic treatment may be included) or solid organ transplantation
* Patients taking at least 2 immunosuppressants
* Patients undergoing combination chemotherapy within the past 3 month 3. One or more of the following:
* Presence of fever at time of screening of ≥ 38.0°C (≥ 100.0°F) taken orally.
* presence of at least one constitutional symptom (headache, myalgia, malaise, or fatigue) of any severity (mild, moderate, or severe),
* presence of at least one respiratory symptoms (e.g. cough, or sore throat) of any severity (mild, moderate, or severe),
* other flu-like symptoms, where the clinician orders a respiratory virus test including influenza A or B 4. Positive test for influenza A (if available) 5. Onset of illness no more than 5 days prior to diagnosis. 6. Females patients of child-bearing age who are capable of conception (i.e. previously have not undergone surgical sterilization) must meet the following criteria:
* Have been sexually abstinent or have used contraceptive agents (oral contraceptive or other hormonal contraceptives including vaginal rings or transdermal patches, intrauterine device (IUD), or barrier methods including condoms) during the 4 weeks prior to date of screening (3 months prior to enrollment for oral/hormonal contraceptives)
* Agree to be sexually abstinent or use contraceptive agents (oral contraceptive or other hormonal contraceptives including vaginal rings or transdermal patches, intrauterine device (IUD), or barrier methods including condoms) from the date of screening through 24 weeks after the last dose of study drug

Exclusion Criteria(all subjects):

1. Nausea that prevents taking oral medications
2. Use of antiviral influenza medication within 10 days(unless switched from randomized to open-label TCAD). An exception to this exclusion criterion may be made by site investigators for patients admitted after hours who receive one or two initial doses of antiviral influenza medication prior to enrollment.
3. Creatinine clearance (estimated by serum creatinine) less than 30 ml/min
4. Current clinical evidence of a recognized or suspected uncontrolled non-influenza infectious illness with onset prior to screening
5. Known hypersensitivity to amantadine, ribavirin, oseltamivir or zanamivir
6. Women who are pregnant (positive serum or urine pregnancy test), who are attempting to become pregnant, or who are breast-feeding
7. Psychiatric or cognitive illness, or recreational drug/alcohol use that, in the opinion of the principal investigator, would affect patient safety and/or compliance
8. Uncontrolled seizure disorder or history of a seizure activity within 12 months prior to study participation
9. Any significant finding in the patient's medical history or physical exam on Day 1 that, in the opinion of the investigator, would affect patient safety or compliance with the dosing schedule
10. Documented Influenza B viral co-infection

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boeckh, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Seattle Children's, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Result] Seo S, Englund JA, Nguyen JT, Pukrittayakamee S, Lindegardh N, Tarning J, Tambyah PA, Renaud C, Went GT, de Jong MD, Boeckh MJ. Combination therapy with amantadine, oseltamivir and ribavirin for influenza A infection: safety and pharmacokinetics. Antivir Ther. 2013;18(3):377-86. doi: 10.3851/IMP2475. Epub 2012 Dec 21. PMID 23264438

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from subjects who had a hematopoietic cell transplantation (HCT) within 2 years or combination chemotherapy within 3 months, those with chronic graft-versus-host disease (GVHD) requiring systemic treatment after 2 years post HCT, or with GVHD taking at least 2 immunosuppressive drugs between February - September, 2009
Groups:
- TCAD; Neuraminidase Inhibitor Monotherapy; Open-labeled TCAD: This substudy was a randomized study comparing a triple combination antiviral drug (TCAD) therapy and oseltamivir (OSL) monotherapy in immunocompromised patients with upper respiratory tract infection due to influenza A who were over 7 years of age and who were not asthmatic.
Period: Overall Study
Arm/Group | TCAD | Neuraminidase Inhibitor Monotherapy | Open-labeled TCAD
Started | 2 | 1 | 4
Completed | 2 | 1 | 3 (One open-labeled patient withdrew on day 5.)
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- TCAD: This substudy was a randomized study comparing TCAD therapy and OSL monotherapy in immunocompromised patients with upper respiratory tract infection due to influenza A who were over 7 years of age and who were not asthmatic.
- Neuraminidase Inhibitor Monotheraphy: Neuraminidase inhibitors include zanamivir and oseltamivir phosphate in this study.
- Open-Labeled TCAD: Subjects with moderate respiratory symptoms and/or influenza-related lower respiratory tract disease, subjects who could not tolerate zanamivir, and children aged 1-6 years received open-label TCAD.
- Total: Total of all reporting groups
Arm/Group | TCAD | Neuraminidase Inhibitor Monotheraphy | Open-Labeled TCAD | Total
Number analyzed (Participants) | 2 | 1 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 2 | 3
  Between 18 and 65 years | 1 | 0 | 2 | 3
  >=65 years | 1 | 0 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 59.5 (17.7) | 17 (0) | 29.5 (26.0) | 36.3 (25.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Drug Specific AEs or AEs Resulting in Treatment Interruption
Description: Abnormal lab data or newly appeared symptoms & signs were considered as AEs.
  Examined lab data:
  Blood cell count (WBC, differential count, Red Blood Cell (RBC), Hemoglobin, Hematocrit, Mean Corpuscular Volume (MCV), Mean Corpuscular Hemoglobin Concentration (MCHC), platelets), Chemistry (Cl, bicarbonate (HCO3), K, Na), Renal function test (BUN, Creatinine, Creatinine clearance), Liver function test (AST, Alanine aminotransferase(ALT), T.Bil, gamma-glutamyltransferase)
Time Frame: 30 days after the final dose of study drug
Measure: Number; unit: number of participants with AEs
Groups:
- TCAD; Open-labeled TCAD: amantadine (75 mg), oseltamivir (50 mg), and ribavirin (200 mg); three times a day for 10 days
- Neuraminidase Inihibitor Monotherapy: oseltamivir (50 mg); three times a day for 10 days
Arm/Group | TCAD | Neuraminidase Inihibitor Monotherapy | Open-labeled TCAD
Number analyzed (Participants) | 2 | 1 | 4
number of participants with AEs | 1 | 1 | 1

2. Secondary Outcome: Number of Participants With Viral Load Decrease as a Function of Time
Description: Viral loads were measured by quantitative Polymerase Chain Reaction (PCR) on day 1, 3, 5, 7, 9, 15, 20 and 28, if applicable.
Time Frame: baseline and 28 days
Population: Three patients could not get viral load at baseline.
Measure: Number; unit: number of participants
Groups:
- TCAD; Neuraminidase Inhibitor Monotherapy: Eligible immunocompromised subjects( age>6 years) positively diagnosed with influenza A who had mild respiratory symptoms were randomized to receive TCAD or neuraminidase inhibitor monotherapy.
- Open-label TCAD: Subjects with moderate respiratory symptoms and/or influenza-related lower respiratory tract disease, subjects who could not tolerate zanamivir, and children aged 1-6 years received.
Arm/Group | TCAD | Neuraminidase Inhibitor Monotherapy | Open-label TCAD
Number analyzed (Participants) | 0 | 1 | 3
number of participants |  | 0 | 2

3. Secondary Outcome: Number of Patients Not Shedding Virus at Day 5 +/-1 and Day 10 +/- 1
Time Frame: 10 days
Population: Participants assessed for viral shedding were those with available baseline viral load data.
Measure: Number; unit: participants
Groups:
- Neuraminidase Inihibitor Monotherapy: Eligible immunocompromised subjects( age>6 years) positively diagnosed with influenza A who had mild respiratory symptoms were randomized to receive TCAD or neuraminidase inhibitor monotherapy.
- Open-labeled TCAD: Subjects with moderate respiratory symptoms and/or influenza-related lower respiratory tract disease, subjects who could not tolerate zanamivir, and children aged 1-6 years received.
Arm/Group | TCAD | Neuraminidase Inihibitor Monotherapy | Open-labeled TCAD
Number analyzed (Participants) | 0 | 1 | 3
participants
  Day 5 +/-1 |  | 0 | 0
  Day 10 +/- 1 |  | 0 | 1

4. Secondary Outcome: Number of Participants With Viral Resistance as a Function of Drug Exposure
Description: Viral resistance was assessed within 28 days after drug administration by detecting resistance-conferring mutation genes and compared to the value at baseline.
Time Frame: 28 days
Population: One open-labeled patient withdrew on day 5.
Measure: Number; unit: Number of participants
Arm/Group | TCAD | Neuraminidase Inihibitor Monotherapy | Open-labeled TCAD
Number analyzed (Participants) | 2 | 1 | 3
Number of participants | 0 | 1 | 0

5. Secondary Outcome: Duration of Symptoms
Description: Calculated as the number of days (mean) any persistent symptom lasted per patient as listed below.
  overall health, short of breath, chills, cough, diarrhea, ear pain, fatigue, fever, headache, hoarseness, muscle ache, phlegm, runny nose, sinus congestion, sneezing, sore throat, watery eyes, wheezing
Time Frame: from baseline up to 28 days
Population: one open labeled patient withdrew on day 5.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TCAD | Neuraminidase Inhibitor Monotherapy | Open-label TCAD
Number analyzed (Participants) | 2 | 1 | 3
days | 4.5 (6.4) | 1 | 4.7 (3.8)

6. Secondary Outcome: Frequency of Confirmed Pneumonia
Time Frame: 58 days
Measure: Number; unit: participants
Arm/Group | TCAD | Neuraminidase Inihibitor Monotherapy | Open-labeled TCAD
Number analyzed (Participants) | 2 | 1 | 4
participants | 0 | 0 | 1

7. Secondary Outcome: Duration of Hospitalization
Time Frame: from baseline up to 58 days
Population: One open-labeled patient withdrew the study on day 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TCAD | Neuraminidase Inihibitor Monotherapy | Open-labeled TCAD
Number analyzed (Participants) | 2 | 1 | 3
days | 6 (8.5) | 6 | 1 (1.7)

8. Secondary Outcome: Days on Supplemental Oxygen
Time Frame: 58 days
Population: One open-labeled TCAD patient withdrew on day 5.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TCAD | Neuraminidase Inihibitor Monotherapy | Open-labeled TCAD
Number analyzed (Participants) | 2 | 1 | 3
days | 2 (1.4) | 0 | 0 (0)

9. Secondary Outcome: Number of Participants With ICU Admissions
Description: The number of participants with ICU admissions was evaluated.
Time Frame: baseline and up to 58 days
Measure: Number; unit: participants
Arm/Group | TCAD | Neuraminidase Inihibitor Monotherapy | Open-labeled TCAD
Number analyzed (Participants) | 2 | 1 | 4
participants | 0 | 0 | 1

10. Secondary Outcome: Number of Participants With Intubations
Time Frame: 58 days
Measure: Number; unit: participants
Arm/Group | TCAD | Neuraminidase Inihibitor Monotherapy | Open-labeled TCAD
Number analyzed (Participants) | 2 | 1 | 4
participants | 0 | 0 | 1

11. Secondary Outcome: Number of Deaths
Time Frame: 58 days
Measure: Number; unit: participants
Groups:
- TCAD: Eligible immunocompromised subjects( age>6 years) positively diagnosed with influenza A who had mild respiratory symptoms were randomized to receiveTCAD or neuraminidase inhibitor monotherapy.
Arm/Group | TCAD | Neuraminidase Inihibitor Monotherapy | Open-labeled TCAD
Number analyzed (Participants) | 2 | 1 | 4
participants | 0 | 0 | 0

12. Secondary Outcome: Pharmacokinetics (AUC0-last) of TCAD
Description: Only 5 patients had partial pharmacokinetic (PK) data available. Plasma concentration of oseltamivir was measured at several time points in one patient receiving neuraminidase inhibitor monotherapy. Plasma concentration of oseltamivir, amantadine, and ribavirin were measured at several time points in four patients receiving TCAD therapy. Area under the time-concentration curve up to the last measured time point (AUC0-last) was calculated from the plasma concentration-time profiles by non-compartmental analysis.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Open-lable TCAD: Subjects with moderate respiratory symptoms and/or influenza-related lower respiratory tract disease, subjects who could not tolerate zanamivir, and children aged 1-6 years received.
Arm/Group | TCAD | Neuraminidase Inhibitor Monotherapy | Open-lable TCAD
Number analyzed (Participants) | 1 | 1 | 3
ng*hr/mL | 304 | 1497 | 2487 (2770)

ADVERSE EVENTS:
Arm/Group | TCAD | Neuraminidase Inihibitor Monotherapy | Open-labeled TCAD
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/1 | 1/4
Other Adverse Events (participants affected / at risk) | 1/2 | 0/1 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCAD (N=2) | Neuraminidase Inihibitor Monotherapy (N=1) | Open-labeled TCAD (N=4)
Acute GVHD (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TCAD (N=2) | Neuraminidase Inihibitor Monotherapy (N=1) | Open-labeled TCAD (N=4)
acute GVHD (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
acute GVHD (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
increased ALP and GGT (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated. Limitations of this study include: small sample size pilot study; inability to enroll the projected number of patients for full analysis before the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes